CLINICAL TRIAL: NCT06213402
Title: A Retrospective/Prospective, Multicenter European Epidemiological Platform for Patients Diagnosed With Rare Anemia Disorders (RADs) With Clinical Significance.
Brief Title: RADeep Multicenter European Epidemiological Platform for Patients Diagnosed With Rare Anemia Disorders (RADs)
Acronym: RADeep
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Erasme University Hospital (Other); Cyprus Institute of Neurology and Genetics (Other); EuroBloodNet Association (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AMI)427/2021
Record Dates: First submitted 2023-12-04; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-12

CONDITIONS: Sickle Cell Disease; Thalassemia; Hemolytic; Anemia, Hereditary, Due to Enzyme Disorder; Anemia Due to Membrane Defect; CDA; Sideroblastic Anemia; Constitutional Aplastic Anemia; Iron Metabolism Disorders; Hereditary Anemia
Keywords: Sickle Cell Disease; Thalassemia; Red Blood Cell; Rare Hematological Disease; Rare Anemia Disorders; Sickle Cell Disease and Related Diseases; Hemoglobinopathy; Beta-Thalassemia; Alpha-Thalassemia; Sickel Cell Anemia; Pyruvate Kinase Deficiency
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Hemolysis; Anemia; Anemia, Sideroblastic; Cystinosis; Iron Metabolism Disorders; Hemoglobinopathies; beta-Thalassemia; alpha-Thalassemia; Pyruvate Kinase Deficiency of Red Cells

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Sickle cell anaemia and other related sickle diseases: Patients with sickle cell disease and related diseases in current regular follow-ups in European-Union health centers
  Interventions: Other: Data collection from EHR.
- Thalassemia and related diseases: Patients with Thalassemia disease and related diseases in current regular follow-ups in European-Union health centers, stratified by age, gender, and/or variants/type if applicable.
  Interventions: Other: Data collection from EHR.
- Pyruvate Kinase Deficiency and related diseases: Patients with Pyruvate Kinase Deficiency and related diseases in current regular follow-ups in European-Union health centers, stratified by age, gender, and/or variants/type if applicable.
  Interventions: Other: Data collection from EHR.
- Red Blood Cell membrane disorders and related diseases: Patients with Reb Blood Cell membrane disorders and related diseases in current regular follow-ups in European-Union health centers, stratified by age, gender, and/or variants/type if applicable.
  Interventions: Other: Data collection from EHR.

INTERVENTIONS:
Other: Data collection from EHR. — Collection of clinical and laboratory data. Reviwe of the electronic health record

SUMMARY:
Rare Anaemia Disorders (RADs) is a group of rare diseases characterized for presenting anaemia as the main clinical manifestation. Different medical entities classified as RADs by ORPHA classification are most of them chronic life threating disorders with many unmet needs for their proper clinical management creating an impact on European health systems. RADs present diagnostic challenges and their appropriate management requires from specialised multidisciplinary teams in Centers of expertise.

Although there are some examples of well-established national registries on RADs in EU, the lack of recommendations for Rare disease registries implementation and the lack of standards for interoperability has led to the fragmentation or unavailability of data on prevalence, survival, main clinical manifestations or treatments in most of the European countries.

DETAILED DESCRIPTION:
The Rare Anaemia Disorders European Epidemiological Platform (RADeep) is an initiative endorsed by the European Reference Network on Rare Hematological Diseases (ERN-EuroBloodNet) under the frame of the European Blood Disorders Platform (ENROL), the ERN-EuroBloodNet umbrella platform officially endorsed by the European Hematology Association (EHA) for European patients' registries on rare haematological diseases. RADeep will share pseudonymised level data with ENROL.

RADeep supports the standardized collection of data of patients affected by any RADs at the European level, maximizing public benefit from data on RADs opened-up with the only restriction needed to guarantee patient rights and confidentiality, in agreement with the General Data Protection Regulation and applicable laws for cross-border sharing of personal data. RADeep has the following major objectives:

1. To collect and describe the demographics, disease-management, and treatment outcomes of patients diagnosed with RADs
2. To perform observational studies concerning research questions and to present outcomes in the fields of health related to organ damage and risk stratification for identification of trial cohorts for new drugs and/or development of research projects
3. To promote harmonization and best practices in the prevention, diagnosis, treatment and follow-up of RADs patients by the dissemination of reliable Guidelines and the translation of research results into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be included in the RADeep Registry
* Age from 0-100, both female and male
* Diagnosed as RADs (SCD, THAL, PKD, and other RADs THAL according to ORPHANET classification)
* Able and willing to provide written informed consent (patient or legal representative for minors)

Exclusion Criteria:

* Patient or legal representative for minors unwilling or unable to give consent
* Patients diagnosed with SCD or THAL (alpha-thalassaemia and beta-thalassaemia) traits or trait conditions for other recessive RADs

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Rade Anemia Disease between 0 - 100 years old that accomplish all the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 32564 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2036-11 (Estimated)

PRIMARY OUTCOMES:
Estimation of Prevalence and Incidence of RADs | 15 years
  Demography and epidemiology
  To collect and to describe demographics and epidemiological data of any type of RADs:
  * Estimate the population frequency of each RAD disease group and disease survival
  * Estimate the diagnosis delay
  * Identify cohorts of patients for research/clinical trials
  * Estimate disease severity
  * Assess the use of specific treatments
  Descriptive analyses will be undertaken at the end of the follow-up period using standard statistical methods to examine the subjects' demographics, disease characteristics and management. Data is updated yearly in an electronic CRF form while assuring homogenization in categorization and units.
  Time-to-event analyses, namely Kaplan-Meier and Cox proportional hazard regression will be used to estimate overall survival.
  Multivariate Cox proportional hazards regression models will be used to identify variables that are important to correlate survival.

CONTACTS AND LOCATIONS:
Overall Officials: María del Mar Manú Pereira, PhD, Principal Investigator — Vall d'hebron Research Institute - Vall d'Hebron Research Institute - University Hospital Vall d'Hebrón (VHIR/HUVH); Béatrice Gulbis, MD, Principal Investigator — Hôpital ERASME (ERASME); Petros Kountouris, PhD, Principal Investigator — Cyprus Institute of Neurology and Genetics (CING)
Locations (1):
- Vall d'hebron Research Institute - Vall d'Hebron Research Institute - University Hospital Vall d'Hebrón (VHIR/HUVH), Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colombatti, R., Gutiérrez-Valle, V., Diot-Lefebvre, C., Labidi, I., Boaro, M.P., Tamana, S., Kountouris, P., Kleanthous, M., Gulbis,B., Mañú-Pereira, M. (2021, October 20). Rare Anaemia Disorders European Epidemiological Platform (RADeep). 17th Annual Sickle Cell & Thalassaemia Conference and 3rd Annual Academy Sickle Cell & Thalassaemia Conference (ASCAT 2022), London, United Kingdom of Great Britain and Northern Ireland.
- See also: EU EurobloodNet offficial Website — https://eurobloodnet.eu/
- See also: RADeep Official Website — https://www.radeepnetwork.eu/
- See also: European Commission website section on European Reference Networks — https://health.ec.europa.eu/european-reference-networks/overview_en

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT06213402/Prot_SAP_000.pdf